CLINICAL TRIAL: NCT03545243
Title: Effect of Proton Pump Inhibitors on the Duodenal Microbiome in Healthy Volunteers and Functional Dyspepsia Patients
Brief Title: PPI and Microbiome in Healthy Volunteers and Functional Dyspepsia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S60984/60953
Record Dates: First submitted 2018-04-24; First posted 2018-06-04 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Dysbiosis
Keywords: duodenum; microbiome; proton pump inhibitor
MeSH Terms: conditions — Dysbiosis | interventions — Pantoprazole

STUDY DESIGN:
Intervention Model Description: Prospective interventional study with study procedures at inclusion, after a baseline period of 4 weeks and Pantoprazole therapy for 4 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pantoprazole 40mg in healthy volunteers (Other): Peroral Pantoprazole 40mg once daily for 4 weeks
  Interventions: Drug: Pantoprazole 40mg
- Pantoprazole 40mg in functional dyspepsia (Other): Peroral Pantoprazole 40mg once daily for 4 weeks
  Interventions: Drug: Pantoprazole 40mg
- PPI-withdrawal in functional dyspepsia (Other): no PPI for 8 weeks
  Interventions: Other: PPI withdrawal

INTERVENTIONS:
Drug: Pantoprazole 40mg — Peroral Pantoprazole 40mg once daily during 28 days
  Other Names: Pantomed
  Arms: Pantoprazole 40mg in functional dyspepsia; Pantoprazole 40mg in healthy volunteers
Other: PPI withdrawal — PPI withdrawal for 8 weeks
  Arms: PPI-withdrawal in functional dyspepsia

SUMMARY:
Prospective interventional study of the effect of PPI on the duodenal microbiome in healthy volunteers and functional dyspepsia patients

DETAILED DESCRIPTION:
PPIs are the first-line therapy in functional dyspepsia (FD) but frequently (over-)prescribed with potential adverse events, especially in the long term. As C. difficile and CAP are important causes of morbidity, mortality and healthcare costs, it is important to study the underlying mechanisms of PPI-induced dysbiosis.

In this prospective interventional study, study procedures will be performed at inclusion (1), after a baseline period of 4 weeks (2) and after treatment with Pantoprazole (Pantomed®) 40mg once daily during 4 weeks (3) in healthy volunteers and FD patients. In addition, study procedures will be performed at inclusion (1) and after PPI-withdrawal for 8 weeks in refractory FD patients.

The investigators aim to assess alterations of the duodenal (mucosa-associated and luminal) microbiome with PPI therapy and to correlate changes in the duodenal microbiota with oral and fecal microbiota, bile acids, intestinal permeability and histology and biochemical variables.

The results from this study will help to unravel the onset and extent of dysbiosis and provide additional arguments not to prescribe or continue PPI without clear clinical indications, especially in cases where alternative regimens may be available or the benefits of PPI are uncertain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 64 years inclusive
* Male or female (not pregnant or lactating and using contraception or postmenopausal)
* Normal bowel habits (defecation once every 3 days up to 3 times a day)
* Witnessed written informed consent
* Access to home freezer (-18 to -20°C)
* Capable to understand and comply with the study requirements

Exclusion Criteria:

* Active psychiatric symptoms (stable dose of single antidepressant allowed)
* Use of acid suppressive drugs (before starting Pantomed), immunosuppressants or antibiotics <3 months before sampling
* Use of drugs influencing stool consistency, NSAIDs, anti-allergy drugs, bile acid sequestrants or ursodeoxycholic acid <2 weeks before sampling
* Use of prokinetics <2 weeks before sampling (unless if ≤3/week)
* History of major abdominal surgery, including cholecystectomy but not appendectomy or splenectomy
* Personal or family (first-degree relative) history of diabetes mellitus type 1, celiac disease, inflammatory bowel disease, psoriasis, rheumatic or other auto-immune diseases (including therapy)
* Allergy or atopy (eczema, asthma and/or allergic rhinoconjunctivitis) (including therapy)
* Kidney, liver or coagulation disorders
* Active coronary or peripheral artery disease
* Diabetes mellitus type 2 (including therapy)
* Active malignancy (including therapy)
* Known HIV, HBV or HCV infection (including therapy)
* Magnetizable objects (e.g. cochlear implants, neural stimulator, pacemaker, metal fragments or implants) or claustrophobia (MRI safety criteria with additional consent form, other procedures can still take place)
* Significant alcohol use (>10 units/weeks)
* Any use of alcohol or smoking ≤2 days before sampling
* Females who are pregnant or lactating, who are not using contraception and premenopausal

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-03-08 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Change in microbiota composition | 4 weeks
  Change in microbiota composition in the duodenum (lumen and mucosa) and feces

SECONDARY OUTCOMES:
Change in mucosal inflammation | 4 weeks
  Change in mucosal inflammation (using immunohistochemistry) of the duodenum
Change in mucosal permeability | 4 weeks
  Change in mucosal permeability (using ussing chambers) of the duodenum
Change in bile acid composition | 4 weeks
  Change in bile acid composition in the duodenum

CONTACTS AND LOCATIONS:
Overall Officials: Tim Vanuytsel, MD PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wauters L, Ceulemans M, Frings D, Lambaerts M, Accarie A, Toth J, Mols R, Augustijns P, De Hertogh G, Van Oudenhove L, Tack J, Vanuytsel T. Proton Pump Inhibitors Reduce Duodenal Eosinophilia, Mast Cells, and Permeability in Patients With Functional Dyspepsia. Gastroenterology. 2021 Apr;160(5):1521-1531.e9. doi: 10.1053/j.gastro.2020.12.016. Epub 2020 Dec 18. PMID 33346007